CLINICAL TRIAL: NCT01014962
Title: A Randomized, Double-Blind, Multiple-Dose, Placebo-Controlled Tolerability And Pharmacokinetic Study Of Escalating Doses Of Albaconazole In Healthy Subjects
Brief Title: A Study of the Effects of Increasing Doses of a Drug for the Treatment of Nail Fungus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 114555
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Onychomycosis
Keywords: Pharmacokinetic; tolerability; multiple escalating doses
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Albaconazole 400 mg cohort 1 (Experimental): Albaconazole 400 mg
  Interventions: Drug: Albaconozole
- Placebo cohort 1 (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo
- Albaconozole 400 mg cohort 2 (Experimental): Albaconozole 400 mg every 12 hours
  Interventions: Drug: Albaconozole
- Placebo cohort 2 (Placebo Comparator): Placebo every 12 hours
  Interventions: Drug: Placebo
- Albaconozole 400 mg cohort 3 (Experimental): Albaconozole 400 mg every 8 hours
  Interventions: Drug: Albaconozole
- Placebo cohort 3 (Placebo Comparator): Placebo every 8 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albaconozole — Albaconozole 400 mg oral once daily for 5 days
  Arms: Albaconazole 400 mg cohort 1
Drug: Placebo — Placebo oral once daily for 5 days
  Arms: Placebo cohort 1
Drug: Albaconozole — Albaconozole 400 mg every 12 hours for 5 days
  Arms: Albaconozole 400 mg cohort 2
Drug: Placebo — Placebo oral every 12 hours for 5 days
  Arms: Placebo cohort 2
Drug: Albaconozole — Albaconozole 400 mg oral every 8 hours for 5 days
  Arms: Albaconozole 400 mg cohort 3
Drug: Placebo — Placebo oral every 8 hours for 5 days
  Arms: Placebo cohort 3

SUMMARY:
The purpose of this study is to determine an upper dose of albaconzole to be administered in a Thorough QTc study.

DETAILED DESCRIPTION:
This study aims to evaluate the safety and tolerability of 5 days of albaconazole dosing at levels that exceed both the projected therapeutic dose and the projected therapeutic frequency, in order to identify an upper dose for administration in a TQTc study. It also aims to assess the pharmacokinetics of multiple escalating doses of albaconazole, and to assess the effects of multiple and sustained dosing of high doses of albaconazole on ECG parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 18 to 45
* A body mass index (BMI) between 18.5 and 30 kg/m2.
* Good physical and mental health.
* Vital signs .within the acceptable range.
* Electrocardiogram (12-lead) after at least 5 minutes in supine position considered as normal or with findings considered as not clinically significant by the investigator. .
* Non-smoker for at least 6 months before screening.
* Subject has screening laboratory parameters within the normal ranges unless considered to be not clinically relevant by the principal investigator. .
* Subject is able to review and understand an informed consent, and must sign the independent ethics committee (IEC)/IRB approved informed consent form before any trial-related procedures are performed.

  * Sexually active females of childbearing potential must have a negative serum pregnancy test result at screening. These subjects must use a medically acceptable method of contraception while receiving protocol-assigned product, and are expected to continue to use this method of contraception for up to 90 days following the last dose of the study medication. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses.

Women who are not currently sexually active or lactating must agree to use 2 forms of nonhormonal contraception, should they become sexually active while participating in the study, and for 90 days following the end of participation in the study. Male subjects and/or their partners must use a medically acceptable form of contraception while receiving protocol-assigned product, and up to 90 days following the last dose of the study medication.

* Subject is willing and able to take the assigned clinical trial medication as directed, comply with clinical trial instructions, and commit to all study visits.

Exclusion Criteria:

* History of intolerance to any of the ingredients in the study medications, or other related drugs, or history of relevant/clinically significant allergic reactions of any origin.
* Any disease or physical condition that, in the opinion of the investigator, could impact the PK/pharmacodynamics of the drug or could potentially compromise the safety of the subject.
* Subject has previously participated in a clinical study of albaconazole.
* History of drug, prescription medicine, or alcohol abuse within the past 2 years.
* Positive drug screen.
* History of psychological or other emotional problems that are likely to invalidate informed consent, or could limit the ability of the subject to comply with the protocol requirements.
* Any drug treatment taken within 14 days before the first drug intake or within 5 half-lives whichever is longer.
* Participation in another clinical trial, blood donation, or significant blood loss less than 30 days before the first intake of study drug.
* Unsuitable veins for repeated venipuncture.
* Subject has any known liver disease or liver toxicity with other drugs.
* Subject has a predose ECG before dosing with a QTcB or QTcF interval >450 msec, or abnormal morphology of the ECG, or clinically serious arrhythmia.
* Subjects who are pregnant, breast-feeding, women of childbearing potential not using adequate contraceptives or planning to conceive, or male subjects who plan to father a child as described in the informed consent.
* Positive for hepatitis B (HBsAg) or hepatitis C (Ab HCV) or HIV or AIDS.
* Consumption of any excluded drugs or foodstuff within 72 hours before dosing.
* Subjects who are employees of a clinical research organization involved in the study, or Stiefel, or an immediate family member.
* Subjects who have a member of the same household in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08-24 (Actual); Primary Completion 2009-12-04 (Actual); Study Completion 2009-12-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of albaconazole in subjects | During 5 days of dosing and 15 days follow-up

SECONDARY OUTCOMES:
Electrocardiogram (ECG) QTc values | During 5 days of dosing and 15 days follow-up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States

REFERENCES:
- See also: Results for study 114555 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114555?search=study&search_terms=114555#rs